CLINICAL TRIAL: NCT04265664
Title: Telerehabilitation With Aims to Improve Lower Extremity Recovery Post-Stroke
Acronym: TRAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Brodie Sakakibara, Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRAIL
Record Dates: First submitted 2020-01-28; First posted 2020-02-11 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Stroke; Stroke, Ischemic; Stroke Hemorrhagic; Cerebral Infarction; Brain Diseases; Central Nervous System Diseases; Cerebral Vascular Disorder; Brain Ischemia; Brain Infarction; Cardiovascular Diseases; Infarction
Keywords: Telerehabilitation; Lower extremity; Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Cerebral Infarction; Brain Diseases; Central Nervous System Diseases; Cerebrovascular Disorders; Brain Ischemia; Brain Infarction; Cardiovascular Diseases; Infarction | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Single-group, pre-post study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation (Experimental): Receives the telerehabilitation protocol
  Interventions: Behavioral: Telerehabilitation

INTERVENTIONS:
Behavioral: Telerehabilitation — Participants in the telerehabilitation program will receive a graded exercise and self-management intervention. This program will be delivered in a ≤2:1 participant:therapist ratio. Each participant grouping will receive two 60-90 minutes telerehabilitation sessions per week for 4 weeks focusing on lower extremity recovery (total 8-12 hours), with a therapist trained in the use of technology for the provision of rehabilitation. Participants will also be asked to complete at least one additional independent self-managed exercise session each week. This independent exercise session will include selected exercises from the telerehabilitation sessions that will be safe to perform without therapist oversight, and jointly agreed upon by the participant and therapist.

SUMMARY:
The purpose of this study is to examine the feasibility and effectiveness of a lower extremity telerehabilitation protocol with aims to improve lower extremity recovery among community-living stroke survivors across Canada.

DETAILED DESCRIPTION:
Eighty percent of stroke survivors experience some form of motor impairment, such as loss or limitation of function in muscle control or movement, or mobility limitation. Regaining walking ability is a priority for most and is achieved in approximately 80%. Unfortunately, the occurrence of falling while walking is as high as 73% of all people who recover the ability to walk post-stroke, with falls often occurring within the first few months of returning home from rehabilitation. This highlights the challenges with transitioning to the community for continued post-stroke rehabilitation. Unfortunately, due to increasing demand on our healthcare and rehabilitation systems and limited service capacity, stroke survivors receive minimal to no follow-up rehabilitation after returning to community-living. As a result, it is common for stroke survivors to report unmet lower extremity rehabilitation needs, and thus ongoing walking/mobility impairment, balance issues, high incidence of falls, and difficulties participating in desired social roles.

The rapid growth in the use of the Internet and personal mobile technologies, including computers, smartphones, and tablets has opened up an array of possibilities through which patients can remotely access specialized health services, such as telerehabilitation supports, while in their homes and communities. The use of technologies to facilitate optimal rehabilitation and recovery after stroke is under-utilized in Canada, despite being highly recommended in Canadian stroke guidelines, and positive beliefs about its potential among people with stroke.

Objectives:

1. To examine the feasibility (e.g. safety, recruitment rate, retention rate, fidelity and adherence, burden) of a lower extremity telerehabilitation protocol among community-living stroke survivors
2. To estimate the size of effect of TRAIL on clinical outcomes of functional mobility, lower extremity strength and motor impairment, functional balance, quality of life, balance self-efficacy, and goal attainment among community-living stroke survivors

Hypotheses:

The investigators expect that the the telerehabilitation protocol will demonstrate sufficient feasibility to support a larger, multisite randomized controlled trial (RCT). The investigators also hypothesize that stroke survivors will improve in functional mobility, lower extremity strength and motor impairment, functional balance, quality of life, balance self-efficacy, and goal attainment following 4-weeks of telerehabilitation with a trained therapist

This feasibility study will use a single group, pre- post- study design trial.

ELIGIBILITY:
Inclusion Criteria:

* 19 year of age or older;
* Within 18 months of the most recent stroke;
* Hemiparesis of the lower extremity;
* Able to walk 10m without physical assistance;
* Able to tolerate 50 minutes of activity (including rest breaks, as needed);
* Have cognitive-communicative ability to participate as per clinical judgement
* Able to provide informed consent;

Exclusion Criteria:

* Currently receiving in- or outpatient rehabilitation;
* Living in long-term care;
* Severe vision or hearing loss;
* Other neurological conditions, e.g. Parkinson's disease;
* Presence of significant comorbidities (e.g. severe osteoarthritis), pain or other symptoms that significantly impact lower extremity function;
* Planned surgery that would preclude or affect participation in the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Timed Up and Go (TUG) at 4 weeks | Baseline, Post-Intervention (immediately following 4 weeks of intervention)
  Performance walking test to assess functional mobility.

SECONDARY OUTCOMES:
Stroke Impact Scale (SIS) | Baseline, Post-Intervention (immediately following 4 weeks of intervention)
  Stroke specific, self-reported health status measure. There are 8 domains assessed in this version and each item is rated using a 5-point Likert scale. The patient rates his/her difficulty completing each item from 1 to 5, and lower scores mean greater difficulty to complete the item.
Activities-Specific Balance (ABC) Scale | Baseline, Post-Intervention (immediately following 4 weeks of intervention)
  Self-reported questionnaire measuring self-efficacy in performing activities without losing balance. The ABC Scale consists of 16 questions that require the patient to rate their confidence on a scale from 0% to 100%. The higher the percentage, the higher level of physical functioning.
Tandem Stand | Baseline, Post-Intervention (immediately following 4 weeks of intervention)
  Performance measure to assess balance through holding a tandem stance position (up to 10 seconds; alternate positions: semi-tandem or feet together).
Functional Reach | Baseline, Post-Intervention (immediately following 4 weeks of intervention)
  Performance measure to assess balance through maximal forward reach (in cm) from a fixed base.
modified virtual Fugl-Meyer Assessment | Baseline, Post-Intervention (immediately following 4 weeks of intervention)
  Performance measure to assess lower extremity impairment.
30 second Sit to Stand | Baseline, Post-Intervention (immediately following 4 weeks of intervention)
  Performance measure used to assess lower extremity strength.
Goal Attainment Scale | Baseline, Post-Intervention (immediately following 4 weeks of intervention)
  An individualized measure involving goal identification, prioritization, and scaling that is standardized to calculate the extent to which a participant's goals are met as a result of the intervention or therapy. Participants rate their goal attainment on a 5-point response scale, ranging from -2 (worse than expected outcome) to +2 (much better outcome), with higher scores indicating a higher degree of goal attainment.

OTHER OUTCOMES:
Feasibility Indicator: Recruitment Rate | Post-Intervention (immediately following 4 weeks of intervention)
  Number of participants recruited.
Feasibility Indicator: Retention Rate | Post-Intervention (immediately following 4 weeks of intervention)
  Percentage of participants with post-intervention data.
Feasibility Indicator: Perceived Benefit of Telerehabilitation | Post-Intervention (immediately following 4 weeks of intervention)
  Satisfaction survey administered at the end of the post-intervention visit.
Feasibility Indicator: Treatment Fidelity | Post-Intervention (immediately following 4 weeks of intervention)
  Percentage of telerehabilitation sessions attended, exercise completed during telerehabilitation sessions, self-managed exercise plans completed.
Feasibility Indicator: Participant Burden | Post-Intervention (immediately following 4 weeks of intervention)
  Percentage of participants with pre- and post-assessments.
Feasibility Indicator: Participant Burden 2 | Post-Intervention (immediately following 4 weeks of intervention)
  Duration to complete the assessments.
Feasibility Indicator: Assessor Burden | Post-Intervention (immediately following 4 weeks of intervention)
  Duration to complete the assessments.
Feasibility Indicator: Therapist Burden | Post-Intervention (immediately following 4 weeks of intervention)
  Time spent administering the telerehabilitation session.
Feasibility Indicator: Ease of Using Equipment | Post-Intervention (immediately following 4 weeks of intervention)
  Downtime due to technical issues of tablet and video-conferencing platform.
Feasibility Indicator: Processing Time | Post-Intervention (immediately following 4 weeks of intervention)
  Time from initial contact to enrolment.
Feasibility Indicator: Incidence of Treatment-Emergent Adverse Events (Safety) | Post-Intervention (immediately following 4 weeks of intervention)
  Adverse events from the telerehabilitation sessions or assessments.
Feasibility Indicator: Treatment Response | Post-Intervention (immediately following 4 weeks of intervention)
  Paired sample t-test.
Feasibility Indicator: Treatment Effect | Post-Intervention (immediately following 4 weeks of intervention)
  Estimate of effect size and variance for future sample size calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Ada Tang, PhD, Principal Investigator — McMaster University; Brodie Sakakibara, PhD, Principal Investigator — University of British Columbia
Locations (5):
- Canada (5):
  - University of British Columbia, Vancouver, British Columbia
  - Riverview Health Centre, Winnipeg, Manitoba
  - Dalhousie University, Halifax, Nova Scotia
  - Parkwood Institute, London, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No